CLINICAL TRIAL: NCT07281339
Title: The Effect of Hypnobreastfeeding Education Given to High-Risk Pregnant Women on Anxiety Levels, Infant Feeding Intention, Postpartum Perception of Insufficient Milk, and Breastfeeding Adaptation
Brief Title: Effect of Hypnobreastfeeding Education in High-Risk Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025000162
Record Dates: First submitted 2025-11-21; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: High-risk Pregnancy; Breast Feeding
Keywords: Hypnobreastfeeding; Anxiety; Infant Feeding Intention; Perception of Insufficient Milk; Breastfeeding Adaptation
MeSH Terms: conditions — Breast Feeding; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Hypnobreastfeeding Education
  Interventions: Behavioral: Hypnobreastfeeding Education
- Control group (No Intervention): Control group

INTERVENTIONS:
Behavioral: Hypnobreastfeeding Education — Monitoring anxiety and breastfeeding intention in pregnancy, and assessing perception of insufficient milk supply, and breastfeeding adaptation in postpartum period
  Arms: Experimental group

SUMMARY:
It is thought that hypnobreastfeeding training given to high-risk pregnant women will reduce anxiety levels, increase lactation, encourage breastfeeding, reduce the perception of insufficient milk, and facilitate adaptation to the postpartum breastfeeding process. According to the results of the power analysis, at least 68 high-risk pregnant women, 34 experimental and 34 control, should be included in the study. Data will be collected with the "Pregnancy Information Form", "Anxiety Assessment Scale", " Infant Feeding Intention Instrument", "Postpartum Information Form", "Perception of Insufficient Milk Questionnaire" and "Breastfeeding Adaptation Scale". In the research, hypnobreastfeeding training will be applied by the researcher to the high-risk pregnant women in the experimental group.

DETAILED DESCRIPTION:
Hypnobreastfeeding training provided to high-risk pregnant women is believed to reduce anxiety, increase lactation, encourage breastfeeding, reduce the perception of insufficient milk supply, and facilitate postpartum breastfeeding adaptation. This will ensure the baby receives adequate and healthy nutrition and the mother's self-confidence increases. Furthermore, hypnobreastfeeding training will contribute to a more comfortable, informed, and peaceful breastfeeding experience for the mother. This will positively impact both the pregnancy and the health of both mother and baby. The study was planned to evaluate the effects of hypnobreastfeeding training given to high-risk pregnant women on anxiety levels, breastfeeding intentions, postpartum perception of insufficient milk, and breastfeeding adaptation. According to the results of the power analysis, at least 68 high-risk pregnant women, 34 experimental and 34 control, should be included in the study. Data will be collected with the "Pregnancy Information Form", "Anxiety Assessment Scale", " Infant Feeding Intention Instrument", "Postpartum Information Form", "Perception of Insufficient Milk Questionnaire" and "Breastfeeding Adaptation Scale". In the research, hypnobreastfeeding training will be applied by the researcher to the high-risk pregnant women in the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* High-risk primiparous pregnant women
* Those with 28-34 weeks of pregnancy
* Those who volunteered to participate in the study
* Those who can read and write Turkish

Exclusion Criteria:

* Those with communication disabilities
* Those with psychiatric and mental illnesses
* Those who have an obstacle to breastfeeding
* Those who have previously attended a birth preparation class
* Those who receive breastfeeding-related training and consultancy
* Those who gave birth prematurely
* Those with anomalies in their babies

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Primiparous high-risk pregnant women
Enrollment: 68 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety Assessment Scale | At the end of the 1 months
  The minimum score that can be obtained from the scale is "10", the maximum score is "50", and as the score obtained from the scale increases, anxiety levels also increase.
Infant Feeding Intention Instrument | At the end of the 1 months
  The minimum score that can be obtained from the scale is "0", the maximum score is "16", and as the score obtained from the scale increases, intention to exclusively breastfeed the baby levels also increase.

SECONDARY OUTCOMES:
Perception of Insufficient Milk Questionnaire | Postpartum 24-48 hours, postpartum 2nd week and postpartum 4th week
  The minimum score that can be obtained from the scale is "0", the maximum score is "50", and as the score obtained from the scale increases, perception of milk sufficiency levels also increase.
Breastfeeding Adaptation Scale | Postpartum 24-48 hours, postpartum 2nd week and postpartum 4th week
  The minimum score that can be obtained from the scale is "27", the maximum score is "135", and as the score obtained from the scale increases, breastfeeding adaptation levels also increase.

CONTACTS AND LOCATIONS:
Overall Officials: Emine İbici Akça, PhD, Principal Investigator — Amasya University
Locations (1):
- Amasya University, Amasya, Turkey (Türkiye)